CLINICAL TRIAL: NCT01163435
Title: Efficacy of High Dose Dual Therapy, Sequential Therapy and Triple Therapy in H. Pylori Eradication - A Prospective, Comparative Study
Brief Title: Efficacy of High Dose Dual Therapy, Sequential Therapy and Triple Therapy in H. Pylori Eradication
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 200912093M
Record Dates: First submitted 2010-07-01; First posted 2010-07-15 (Estimated); Last update posted 2013-12-03 (Estimated); Status verified 2013-12

CONDITIONS: Helicobacter Infection
Keywords: Helicobacter pylori; antibiotic resistance; high dose dual therapy; sequential therapy; clarithromycin-based triple therapy; levofloxacin-based triple therapy
MeSH Terms: conditions — Helicobacter Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- high dose dual therapy (Experimental): group A1 and A2 - high dose dual therapy (rabeprazole 20 mg qid, amoxicillin 750 mg qid for 14 days)
  Interventions: Drug: high dose dual therapy
- sequential therapy (Experimental): group B1 and B2 - sequential therapy (rabeprazole 20 mg, amoxicillin 1000 mg, bid for 5 days, then rabeprazole 20 mg , metronidazole 500 mg, clarithromycin 500 mg, bid for next 5 days)
  Interventions: Drug: sequential therapy
- clarithromycin-based triple therapy (Active Comparator): group C1 - clarithromycin-based triple therapy (rabeprazole 20 mg, amoxicillin 1000 mg, clarithromycin 500 mg, bid for 7 days)
  Interventions: Drug: clarithromycin-based triple therapy
- levofloxacin-based triple therapy (Active Comparator): group C2 - levofloxacin-based triple therapy (rabeprazole 20 mg, amoxicillin 1000 mg, levofloxacin 250 mg, bid for 7 days)
  Interventions: Drug: levofloxacin-based triple therapy

INTERVENTIONS:
Drug: high dose dual therapy — rabeprazole 20 mg qid,amoxicillin 750 mg qid for 14 days
  Arms: high dose dual therapy
Drug: sequential therapy — rabeprazole 20 mg, amoxicillin 1000 mg, bid for 5 days, then rabeprazole 20 mg , metronidazole 500 mg, clarithromycin 500 mg, bid for next 5 days
  Arms: sequential therapy
Drug: clarithromycin-based triple therapy — rabeprazole 20 mg, amoxicillin 1000 mg, clarithromycin 500 mg, bid for 7 days
  Arms: clarithromycin-based triple therapy
Drug: levofloxacin-based triple therapy — rabeprazole 20 mg, amoxicillin 1000 mg, levofloxacin 250 mg, bid for 7 days
  Arms: levofloxacin-based triple therapy

SUMMARY:
Up to now, to our knowledge, there is few randomized, large scale study prospectively and simultaneously comparing the efficacy, adverse effects and patient adherence of these current recommended 1st-line or 2nd-line regimens for H. pylori eradication in and out of our country.

The aims of this study are:

1. to compare the efficacy of high dose dual therapy, sequential therapy and clarithromycin-based triple therapy as 1st-line regimen in H. pylori eradication;
2. to compare the efficacy of high dose dual therapy, sequential therapy and levofloxacin-based triple therapy as rescue regimen in H. pylori eradication;
3. to compare the patient adherence and adverse effects of these treatment regimens;
4. to investigate factors that may influence H. pylori eradication by these treatment regimens;
5. to investigate and analyze the prevalence and trend of antibiotic resistance.

DETAILED DESCRIPTION:
Patients having H. pylori-positive chronic gastritis with/without peptic ulcers will be recruited. All undergo endoscopy with biopsy before treatment. Four to eight weeks after termination of treatment, H. pylori infection status will be examined by endoscopy with biopsy or the Carbon 13-urea breath test if the patients refuse the second endoscopy. The cytochrome P450 (CYP) 2C19 genotype of each participant will be analyzed by the polymerase chain reaction-based restriction fragment length polymorphism (PCR-RFLP) method. A computed generated random numbers sequence will be blocked into three subgroups, say A1, B1 and C1 (or A2, B2, and C2).

If the patients did not receive anti-H. pylori therapy previously, they will be invited to enter the first part of study for evaluating the efficacy of 1st-line regimens. If the patients had received anti-H. pylori therapy previously, they will be invited to enter the second part of study for evaluating the efficacy of rescue regimens. Patients who meet the inclusion criteria and do not have any one of the exclusion criteria will be randomized to receive one of the following regimens:

* for 1st-line regimens: group A1 - high dose dual therapy (rabeprazole 20 mg qid + amoxicillin 750 mg qid for 14 days); group B1 - sequential therapy (rabeprazole 20 mg + amoxicillin 1000 mg, bid for 5 days, then rabeprazole 20 mg + metronidazole 500 mg + clarithromycin 500 mg, bid for next 5 days); group C1 - clarithromycin-based triple therapy (rabeprazole 20 mg + amoxicillin 1000 mg + clarithromycin 500 mg, bid for 7 days).
* for rescue regimens: group A2 - high dose dual therapy (as group A1); group B2 - sequential therapy (as group B1); group C2 - levofloxacin-based triple therapy (rabeprazole 20 mg + amoxicillin 1000 mg + levofloxacin 250 mg, bid for 7 days).

All patients will be asked to complete a questionnaire and to record symptoms and drug consumption daily during the treatment period. Post-treatment, the patients were seen at the Outpatients Clinic to investigate patient adherence and adverse effects of treatment.

ELIGIBILITY:
Inclusion Criteria:

* patients having H. pylori related chronic gastritis with/without peptic ulcers who are aged greater than 18 years and are willing to received eradication therapy.

Exclusion Criteria:

* pregnant or nursing woman
* serious concomitant illness and malignant tumor of any kind
* history of hypersensitivity to test drugs
* serious bleeding during the course of this ulcer
* previous gastric surgery
* receiving bismuth salts, proton pump inhibitors, or antibiotics in the previous month.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 618 (Actual)
Dates: Start 2010-08; Primary Completion 2013-07 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
to compare the efficacy, adverse effects and patient adherence of high dose dual therapy, sequential therapy and clarithromycin-based triple therapy (or levofloxacin-based triple therapy) as 1st-line regimen (or rescue regimen) in H. pylori eradication | 3.5 years
  The eradication rates (efficacy) will be evaluated by intention-to-treat (ITT) and per-protocol (PP) analysis. The safety and tolerability will be evaluated by the number of participant with adverse events and patient adherence (by counting unused medication after the treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Jyh-Chin Yang, M.D.Ph.D., Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Yang JC, Lin CJ, Wang HL, Chen JD, Kao JY, Shun CT, Lu CW, Lin BR, Shieh MJ, Chang MC, Chang YT, Wei SC, Lin LC, Yeh WC, Kuo JS, Tung CC, Leong YL, Wang TH, Wong JM. High-dose dual therapy is superior to standard first-line or rescue therapy for Helicobacter pylori infection. Clin Gastroenterol Hepatol. 2015 May;13(5):895-905.e5. doi: 10.1016/j.cgh.2014.10.036. Epub 2014 Nov 14. PMID 25460556